CLINICAL TRIAL: NCT02218736
Title: A Phase 2a Study to Evaluate the Kappa Opioid Receptor As a Target for the Treatment of Mood and Anxiety Spectrum Disorders by Evaluation of Whether CERC-501 Engages Key Neural Circuitry Related to the Hedonic Response
Brief Title: Fast-Fail Trials in Mood and Anxiety Spectrum Disorders; Kappa Opioid Receptor Phase 2a
Acronym: FASTMAS_Kor2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Yale University (Other); Baylor College of Medicine (Other); Indiana University (Other); Icahn School of Medicine at Mount Sinai (Other); Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: Pro00052485; HHSN271201200006I (Other: NIH/NIMH)
Record Dates: First submitted 2014-08-15; First posted 2014-08-18 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: ANXIETY DISORDERS (or Anxiety and Phobic Neuroses)
Keywords: Anhedonia; Mood and Anxiety Spectrum Disorders; CERC-501 (investigational product); Kappa Opioid Receptor (KOR)
MeSH Terms: conditions — Anxiety Disorders; Phobic Disorders; Anhedonia | interventions — Aticaprant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CERC-501 (Experimental): Oral dosing of 10 mg CERC-501 (formerly known as LY2456302) administered daily for 8 weeks
  Interventions: Drug: CERC-501
- Placebo (Placebo Comparator): Oral daily administration of 10 mg placebo for 8 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: CERC-501 — Oral dosing of 10 mg CERC-501 daily for 8 weeks
  Other Names: Kappa Opioid Receptor Antagonist; LY2456302
  Arms: CERC-501
Drug: placebo — oral dosing of 10 mg placebo daily for 8 weeks
  Arms: Placebo

SUMMARY:
The available treatment for patients with mood and anxiety disorders have significant limitations (Rush, 2007; Denys and de Geus, 2005). There is a need to develop new treatments for people with these disorders. Many research studies carried out in animals and a few preliminary studies carried out in humans suggest that medications which block kappa opioid receptors (KOR) have potential for being effective new treatments for patients with mood and anxiety spectrum disorders. These medications have shown particular promise for improving one important type of difficulty experienced by many patients who suffer from mood and anxiety spectrum disorders referred to as anhedonia, which is an impairment in reward-related function. In this study we will test the hypothesis that KOR antagonism is a promising means of improving anhedonia in patients with mood and anxiety spectrum disorders. We will do so by evaluating whether we can establish Proof of Concept (POC) that a relatively selective KOR antagonist, CERC-501 (formerly known as LY2456302), engages neural circuits involved in mediating reward-related function in patients with mood and anxiety spectrum disorders with anhedonia. We are attempting to establish POC in this study in order to determine whether there is a sufficient basis for pursuing future work evaluating whether KOR antagonism has therapeutic effects on clinical and behavioral measures of reward-related functioning.

DETAILED DESCRIPTION:
FAST-MAS addresses an important problem and critical barrier to progress in Mood and Anxiety Spectrum Disorders and if the aims of the project are achieved, FAST-MAS could shift scientific knowledge, technical capacity, and clinical practice in a positive direction.

The Mood and Anxiety Spectrum disorders are both extremely common and associated with significant morbidity and mortality and, as such, represent an important public health problem in the United States.

The mood disorders include the following diagnostic entities: major depressive disorder (MDD), bipolar disorder (including subtypes of mania, mixed state, and depressed, as well as types I and II), and dysthymic disorder. Available epidemiologic data suggest that the prevalence of these mood disorders is extremely high among adults in the United States, approaching 10%. Among the mood disorders, MDD has high lifetime prevalence, with recent estimates up to 16%. According to the World Health Organization (WHO), MDD is currently the leading cause of disability with the greatest burden of illness in developed countries and the third most common cause of disability worldwide. MDD is life shortening due to both suicide and its association with increased mortality from other medical conditions. It is also a highly recurrent condition with between 50% and 75% of persons diagnosed with MDD experiencing more than one episode. Bipolar Disorder is also a highly recurrent condition. The lifetime prevalence of bipolar disorder has been estimated to be approximately 3.4% in the World Health Survey Initiative. Approximately 60% of affected individuals experience severe or very severe role impairment based on the Sheehan Disability Scale and, like MDD, bipolar disorder is associated with significant suicide risk.

The anxiety disorders are also very common and associated with significant adverse impact on affected individuals and society. These disorders include the following diagnostic entities: generalized anxiety disorder (GAD), panic disorder, obsessive-compulsive disorder, social phobia, specific phobias, and post-traumatic stress disorder (PTSD). As a group, these conditions affect approximately 18% of adults in a given year and they are associated with significant co-morbidities and adverse consequences. Of the anxiety disorders, GAD appears to be associated with the greatest per patient cost and disability with a degree of disability comparable to that of MDD and comparable to chronic medical conditions such as arthritis, diabetes, and peptic ulcer disease. It affects approximately 6.8 million adults in the U.S. and is a highly chronic condition. Panic disorder affects about 6 million American adults and is twice as common in women as men. Panic disorder is also highly disabling and often chronic and even mild forms of this disorder are linked to significantly increased impairment in function and quality of life as well as a number of comorbidities. Approximately 2.2 million adults in the U.S. are affected by obsessive-compulsive disorder and this disorder is often accompanied by psychiatric comorbidities. Roughly half of individuals with this condition have a chronic unremitting course which is associated with significant disability and morbidity. Social phobia, also known as social anxiety disorder, is seen in roughly 15 million adults in the U.S. and is often associated with MDD or other anxiety disorders. It is generally a chronic condition that leads to a great degree of disability due to substantial impairment in social, educational, and occupational function. Approximately 8 million adults in the U.S. experience PTSD and approximately 12% of the population have PTSD at some point in their lives and affected individuals frequently experience associated MDD, other anxiety disorders and substance use problems. The level of disability associated with this condition tends to be quite high and includes impairment in social and occupational function and quality of life. There are also substantial financial and social costs associated with PTSD due to increased hospitalization rates, suicidality, and substance use problem.

Mood disorders and anxiety disorders are highly prevalent conditions, many of which are chronic, nearly all of which are associated with substantial comorbidities, disability and impairment and some are associated with an increased risk for mortality. Despite the availability of many pharmacologic, psychotherapeutic, brain stimulation, and combination treatment options available to clinicians, many patients with Mood and Anxiety Spectrum Disorders respond poorly to treatment. In light of the impairments, costs, and risks of these disorders, the limitations of the available treatments represents an enormous burden to public health and speak strongly to the need for new treatments for these conditions as well as novel methodologies of treatment development that are not only faster than existing methodologies but which also promote new ways of thinking about these disorders and their treatment and capitalize on recent and ongoing developments in basic science.

This study will be a six-site randomized, double-blind, PBO (placebo) -controlled, parallel-group mono-therapy study to assess the effects of CERC-501 (formerly known as LY2456302) compared to PBO in adults age 21-65 years with mood and anxiety spectrum disorders. We will recruit a total of 90 subjects, of which 45 will be randomized to CERC-501 and 45 to placebo for 8 weeks of treatment

ELIGIBILITY:
Inclusion Criteria:

* Age between 21 and 65 years of age
* Must meet DSM-IV TR (Diagnostic and Statistical Manual of Mental Disorders, 4th edition, text revision) diagnostic criteria for: Major Depressive Disorder, Bipolar I or II Depressed, Generalized Anxiety Disorder, Social Phobia, Panic Disorder, or Post Traumatic Stress Disorder
* Snaith-Hamilton Pleasure Scale (SHAPS) score ≥ 20
* Reliable and willing to be available for the duration of the study
* Willing and able to give written informed consent to participate
* Able to understand and comply with instructions
* If female of childbearing potential, must agree to use dual methods of contraception and be willing and able to continue contraception for 6 weeks after the last dose of study drug. Females using oral contraception must have started using it at least 2 months prior to the Baseline Visit
* If male of childbearing potential, must have undergone surgical sterilization (such as a vasectomy) or agree to use a condom used with a spermicide during participation in the study and for 1 month afterward

Exclusion Criteria:

* Expected to require hospitalization during the course of the study
* Current/history of a psychotic disorder, current manic or mixed episode, autism spectrum disorders, mental retardation
* Met DSMIV-TR (Diagnostic and Statistical Manual of Mental Disorders, 4th edition, text revision) criteria for substance abuse within the last 3 months or substance dependence within the last 6 months, excluding caffeine and/or nicotine
* History of unstable or untreated serious medical condition based on physician evaluation, medical history, and screening laboratory testing
* Active suicidal intent or plan, or history of attempt within the past 3 months based on physician evaluation and Columbia Suicide Severity Rating Scale (C-SSRS)
* Use of any antidepressant, antipsychotic, anxiolytic, anticonvulsant, mood stabilizing, muscle relaxant, centrally acting antihistaminergic, stimulant or insomnia medications (See Appendix 2) within 5 half-lives of baseline or at any time during after baseline
* Use of any medication that is primarily metabolized by Cytochrome P450 2C8 within 14 days of baseline or at any time during the study. This includes: Cerivastatin, Paclitaxel, Repaglinide, Sorafenib, Rosiglitazone, Trimethoprim, Amodiaquine, Morphine, Amiodarone, Cabazitaxel, Carbamazepine, Chloroquine, Ibuprofen, Trepostinil, Torsemide.
* Any contraindications to the magnetic resonance imaging procedures
* Positive urine drug screen at any time during the study
* Use of any investigational medication within 3 months prior to the start of this study or scheduled to receive an investigational drug other than the study drug during the course of this study
* Known hypersensitivity to CERC-501 (formerly known as LY2456302)
* History of severe allergies or multiple adverse drug reactions
* History of gastric disease (including peptic ulcer disease, gastritis, upper GI bleeding, or any GI precancerous condition), current clinically evident gastrointestinal complaints, or positive urea breath test
* Current use of a proton pump inhibitor or histamine 2 blocker, or a history of chronic NSAID (nonsteroidal anti-inflammatory drug) use.
* History of use of Salvia divinorum or use of Salvia divinorum at any time during the study.
* Any other condition that in the opinion of the investigator would preclude participation in the study
* Any smoking of cigarettes or use of other nicotine containing products within the last month or at any time during the study
* Pregnant or lactating

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Weiner, MD, PhD, Principal Investigator — Duke University
Locations (6):
- United States (6):
  - Yale University, New Haven, Connecticut
  - Andrew Goddard, MD, Indianapolis, Indiana
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - CaseWestern Reserve University, Cleveland, Ohio
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Background] Rorick-Kehn LM, Witkin JM, Statnick MA, Eberle EL, McKinzie JH, Kahl SD, Forster BM, Wong CJ, Li X, Crile RS, Shaw DB, Sahr AE, Adams BL, Quimby SJ, Diaz N, Jimenez A, Pedregal C, Mitch CH, Knopp KL, Anderson WH, Cramer JW, McKinzie DL. LY2456302 is a novel, potent, orally-bioavailable small molecule kappa-selective antagonist with activity in animal models predictive of efficacy in mood and addictive disorders. Neuropharmacology. 2014 Feb;77:131-44. doi: 10.1016/j.neuropharm.2013.09.021. Epub 2013 Sep 23. PMID 24071566

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 69 participants screen failed, 2 were unable to complete baseline per protocol, 3 withdrew consent prior to baseline.
Period: Overall Study
Arm/Group | CERC-501 | Placebo
Started | 45 | 44
Completed | 33 | 35
Not Completed | 12 | 9
Not completed — Withdrawal by Subject | 10 | 9
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Population: Participants who were randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | CERC-501 | Placebo | Total
Number analyzed (Participants) | 45 | 44 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 44 | 89
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (13.30) | 38.2 (13.02) | 39.5 (13.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 27 | 56
  Male | 16 | 17 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 38 | 38 | 76
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 8 | 18
  White | 31 | 28 | 59
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45 | 44 | 89

OUTCOME MEASURES:

1. Primary Outcome: Change in Ventral Striatal Activation Occurring in Anticipation of Reward During the Monetary Incentive Delay Task Measured by fMRI
Description: Establish POC (Proof of Concept) for KOR (Kappa Opioid Receptor) antagonism by evaluating the impact of CERC-501 relative to Placebo on reward-related neural circuitry in terms of ventral striatal activation during anticipation of reward during the Monetary Incentive Delay Task. Evaluation by fMRI (Functional magnetic resonance imaging). The BOLD (Blood Oxygen Level-Dependent) score on the Z-scale represents how far the actual measured intensity is from the expected in the template. A score of 0 would correspond to the mean/median, a score of 1.65 would represent the 90-percentile, -1.65 the 10-percentile, and so on, according to a standard normal distribution.
Time Frame: baseline, Week 8
Population: The primary and secondary endpoints are analyzed for patients who meet the definition of completers for week 8 of the study.
Measure: Mean (95% Confidence Interval); unit: Z score
Arm/Group | CERC-501 | Placebo
Number analyzed (Participants) | 34 | 34
Z score | 0.718 [0.487 to 0.950] | 0.331 [0.103 to 0.559]
Statistical Analysis 1: Comparison: CERC-501 vs Placebo; Test type: Superiority; p = 0.0095, t-test, 1 sided

2. Secondary Outcome: Clinical Anhedonia Measured by the Snaith-Hamilton Pleasure Scale (SHAPS; Total Score)
Description: To determine if CERC-501 is superior to placebo in improving a clinical self-report measure of anhedonia using the Snaith Hamilton Pleasure Scale (SHAPS). A single value was calculated for the average over 8 weeks. The SHAPS is a well-validated 14-item questionnaire used to assess anhedonia. It asks participants to agree or disagree with statements of hedonic response in pleasurable situations. Four responses are possible: Strongly disagree, Disagree, Agree, or Strongly agree. Each item is worded so that higher scores indicate greater pleasure capacity. A total score is derived by summing the responses to each item. Items answered "strongly agree" are coded as "1", while "strongly disagree" are coded a score of "4." Therefore, scores on the SHAPS can range from 14 to 56, with higher scores corresponding to higher levels of anhedonia.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CERC-501 | Placebo
Number analyzed (Participants) | 34 | 34
score on a scale | 30.777 [29.547 to 32.007] | 32.363 [31.157 to 33.568]
Statistical Analysis 1: Comparison: CERC-501 vs Placebo; Test type: Superiority; p = 0.0345, t-test, 1 sided

3. Secondary Outcome: Change in Behavioral Measure of Anhedonia Using the Probabilistic Reward Task
Description: To evaluate the impact of CERC-501 relative to placebo on a behavioral measure of anhedonia using the Probabilistic Reward Task (PRT). The PRT will be carried out at baseline and after 8 weeks of double-blind treatment to assess the effects on a behavioral outcome measure that assessed reward-related function (level of reward learning). The score obtained is a ratio of the number of times participants correctly choose the high reward stimuli versus the low rewarding stimuli
Time Frame: baseline, Week 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Ratio (Response Bias Score)
Arm/Group | CERC-501 | Placebo
Number analyzed (Participants) | 34 | 34
Ratio (Response Bias Score) | 0.034 [-0.019 to 0.087] | 0.019 [-0.030 to 0.068]
Statistical Analysis 1: Comparison: CERC-501 vs Placebo; Test type: Superiority; p = 0.430, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of consent through 12 weeks for all subjects.
Arm/Group | CERC-501 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/44
Other Adverse Events (participants affected / at risk) | 34/45 | 32/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CERC-501 (N=45) | Placebo (N=44)
Diarrhea (Gastrointestinal disorders) | 13 | 8
Headache (Nervous system disorders) | 10 | 10
Suicidal Ideation (Psychiatric disorders) | 9 | 7
Puritus (Skin and subcutaneous tissue disorders) | 10 | 2
Depression (Psychiatric disorders) | 6 | 5
Dizziness (Nervous system disorders) | 6 | 5
Anxiety (Psychiatric disorders) | 6 | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 4 | 5
Dry Mouth (Gastrointestinal disorders) | 4 | 4
Insomnia (Nervous system disorders) | 4 | 4
Nausea (Gastrointestinal disorders) | 3 | 5
Pollakiuria (Renal and urinary disorders) | 4 | 3
Rash (Skin and subcutaneous tissue disorders) | 6 | 1
Constipation (Gastrointestinal disorders) | 4 | 1
Fatigue (General disorders) | 3 | 2
Tinnitus (Ear and labyrinth disorders) | 4 | 1
Vission Blurred (Eye disorders) | 4 | 1
Coordination Abnormal (Nervous system disorders) | 3 | 1
Disturbance in Attention (Psychiatric disorders) | 3 | 1
Dizziness postural (Nervous system disorders) | 3 | 1
Non-cardiac chest pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Restlessness (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Dysuria (Renal and urinary disorders) | 3 | 0
Hyperhidrosis (General disorders) | 2 | 1
Hypersomnia (Psychiatric disorders) | 1 | 2
Irritability (General disorders) | 2 | 1
Libido decreased (Reproductive system and breast disorders) | 1 | 2
Asthenia (General disorders) | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Malaise (General disorders) | 2 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 2
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Palpitations (Cardiac disorders) | 0 | 2
Panic attack (Nervous system disorders) | 1 | 1
Pyrexia (General disorders) | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1
Anal pruritus (Gastrointestinal disorders) | 1 | 0
Blepharitis (Eye disorders) | 1 | 0
Chest discomfort (Cardiac disorders) | 1 | 0
Chest pain (Cardiac disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Depressive symptom (Psychiatric disorders) | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 0
Initial insomnia (Psychiatric disorders) | 1 | 0
Intentional self-injury (Psychiatric disorders) | 0 | 1
Middle insomnia (Psychiatric disorders) | 0 | 1
Mood altered (Psychiatric disorders) | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Night sweats (General disorders) | 0 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1
Sedation (Nervous system disorders) | 0 | 1
Self-injurious ideation (Psychiatric disorders) | 1 | 0
Syncope (Vascular disorders) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Tension headache (Nervous system disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Urinary track infeciton (Renal and urinary disorders) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-10-06): https://cdn.clinicaltrials.gov/large-docs/36/NCT02218736/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/36/NCT02218736/SAP_001.pdf